CLINICAL TRIAL: NCT01876888
Title: Turkish Version of MedRisk Instrument for Measuring Patient Satisfaction With Physical Therapy Care: Its Cultural Adaptation, Validation and Reliability Study
Brief Title: Turkish Cultural Adaptation, Validation and Reliability Study of MedRisk Instrument
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Cigdem Ayhan, Lecturer, Hacettepe University
Other Study IDs: Physiotherapy & Rehabilitation
Record Dates: First submitted 2013-06-07; First posted 2013-06-13 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Cultural Adaptation
Keywords: patient satisfaction; physical therapy; MedRisk instrument
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
The aims of this study were to perform cultural adaptation of the MedRisk Instrument for Measuring Patient Satisfaction With Physical Therapy Care (MRPS) instrument and provide information regarding the factor structure, group-level reliability, and criterion-referenced validity of the instrument in Turkish speaking patients.

DETAILED DESCRIPTION:
Patient satisfaction with physical therapy has become an important concern in health care, used to monitor patient perceptions of the quality of physical therapy care services. Measurement of patient satisfaction may provide useful information which may improve the quality of health care. The "MedRisk Instrument for Measuring Patient Satisfaction With Physical Therapy Care" (MRPS) is one of these instruments, which has undergone reliability and validation testing.The MRPS is a 20-item (18 items and 2 global measures) questionnaire which assess patient experience about therapist, registration process and convenience of environment.

A survey on a consecutive sample of patients from various regions in Turkey who were receiving outpatient physiotherapy programs was recruited.The study was divided into two phases: Phase I, the cross-cultural adaptation, which involves the translation procedures into Turkish and preliminary probe in the target population; and phase II, which involves the reliability and validation study.

After providing informed consent, for test-retest reliability, all subjects were asked to complete the MRPS twice; the first at least after receiving three sessions of physiotherapy and the second four days later which could coincide with the date of their discharge but not later. Subjects provided information regarding their age, sex, and location of primary symptoms prior to completing the instrument.Factor structure.

The construct validity was evaluated by factor analysis method. An exploratory factor analysis, using principal components analysis with varimax rotation was performed.Criterion validity was addressed by determining the correlation between two global measures of satisfaction and each of the 18 items. The measurement properties of the potential factors were investigated by determining correlations of the factors to the global measures and 10-cm Visual Analog Scale (VAS) which evaluates the level of patient satisfaction with higher scores indicating better satisfaction. Pearson correlation coefficient was used to assess the strength of the linear relationships. Test-retest reliability was examined by calculating the Intraclass Correlation Coefficient (ICC). Internal consistency relates to homogeneity of an instrument, which is assessed with Cronbach's alpha

ELIGIBILITY:
Inclusion Criteria:

* All subjects had to be able to read and write in Turkish.

Exclusion Criteria:

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from various regions in Turkey who were receiving outpatient physiotherapy programs.
Sampling Method: Non-Probability Sample
Enrollment: 317 (Actual)
Dates: Start 2011-04; Primary Completion 2012-09 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
patient satisfaction instrument | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Özgen Aras, Study Director — T.C. Dumlupınar Üniversitesi; Cigdem Ayhan, Principal Investigator — Hacettepe University; Yavuz Yakut, Study Chair — Hacettepe University